CLINICAL TRIAL: NCT02908945
Title: The Effect of Ketamine on the WAVCNS Index During General Anesthesia: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Richard Merchant, Anesthesiologist, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHREB 2016-054
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Anesthesia
Keywords: Ketamine; Anesthesia; EEG; NeuroSENSE; Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Participants randomized to group 1 will receive a 0.5 mg/kg loading dose of racemic ketamine hydrochloride immediately before induction of anesthesia, followed by a continuous 10 mcg/kg/min infusion throughout maintenance of anesthesia, until procedure end (last suture inserted), up to a maximum cumulative dose of 200 mg. Participants will recieve EEG monitoring with the NeuroSENSE monitor.
  Interventions: Drug: Ketamine; Device: NeuroSENSE monitor
- Group 2 (Experimental): Participants randomized to group 2 will receive a 0.25 mg/kg loading dose of racemic ketamine hydrochloride immediately before induction of anesthesia, followed by a continuous 5 mcg/kg/min infusion throughout maintenance of anesthesia, until procedure end (last suture inserted), up to a maximum cumulative dose of 200 mg. Participants will recieve EEG monitoring with the NeuroSENSE monitor.
  Interventions: Drug: Ketamine; Device: NeuroSENSE monitor
- Group 3 (Other): Participants randomized to the control group will receive an equivalent anesthetic, without the addition of ketamine. Participants will recieve EEG monitoring with the NeuroSENSE monitor.
  Interventions: Device: NeuroSENSE monitor

INTERVENTIONS:
Drug: Ketamine — Bolus dose before induction of anesthesia and infusion during maintenance of anesthesia.
  Other Names: Ketalar
  Arms: Group 1; Group 2
Device: NeuroSENSE monitor — NeuroSENSE monitors the brain using electroencephalography (EEG) and produces an index called the WAVCNS. WAVCNS is a measure of depth of hypnosis (DoH).

SUMMARY:
Monitoring the brain using electroencephalography (EEG) during general anesthesia provides the anesthesiologist with valuable feedback of how deeply anesthetized their patient is, reducing the chances of under- or overdosing and potentially improving patient outcomes. However, commercial EEG monitors that output processed EEG (pEEG) were developed under carefully controlled, simple anesthetic regimes - in contrast to the multimodal "cocktail" of drugs often used in clinical practice. Ketamine is one potential adjunct to a standard anesthetic, which has a growing body of evidence suggesting that it may improve post-operative outcomes. The effects of ketamine on pEEG parameters are poorly understood. This randomized, open-label, feasibility study will be undertaken in a sample of 30 adult outpatient surgery patients. The primary objective is to observe the intra-operative raw and pEEG trends using the NeuroSENSE monitoring system in patients receiving one of two different analgesic doses of ketamine, compared to patients not receiving ketamine, during an otherwise comparable general anesthetic. Secondarily, we will consider other clinical data of interest from both intra- and post-operative contexts in order to establish a broader understanding of the potential influence of two analgesic ketamine doses on anesthetic depth and post-operative outcomes. Feasibility outcomes will be assessed with the ultimate goal of developing a larger-scale clinical trial.

DETAILED DESCRIPTION:
Purpose of Study The primary aim of this study is to analyze the effect of two different intra-operative ketamine doses, within the low, analgesic range, on raw and processed EEG (the WAVCNS) during induction, maintenance, and emergence from general anesthesia compared to a no-ketamine control group. These data will be compared against other more traditional measures of depth of hypnosis (DoH), such as drug requirements, blood pressure, heart rate, and the occurrence of any unwanted intra-operative events. Ultimately, the results of this study will be used to assess whether or not it is feasible to rely on the WAVCNS index, as a valid measure of anesthetic effect, when either of these doses of ketamine has been added to an anesthetic regime. This will inform the feasibility of a larger trial comparing the effect of low dose ketamine on the performance of an automated anesthesia system.

Secondarily, this study aims to observe certain post-operative outcomes that have previously been shown to be influenced by ketamine administration, in order to better understand the potential for patient benefit associated with these doses of ketamine. Specifically, we will record pain intensity, opioid requirements, PONV, dreaming, and shivering occurring in the post-anesthesia care unit (PACU).

Justification for Study The amount of anesthetic required to maintain an adequate DoH varies widely between individual patients, and within patients under different conditions. Processed EEG-based DoH monitors provide the opportunity to deliver drugs at a dose more appropriate to a patient according to dynamic feedback of therapeutic effect. As a result, the quality of an anesthetic regimen and patient outcomes may be improved. However, since pEEG values are affected differently by different types and doses of drugs, these monitors would be much better utilized if the effects of certain drugs on processed values were better defined. Accumulating evidence suggests that the use of low dose intra-operative ketamine has the potential to be clinically beneficial, especially in terms of reducing post-operative pain, which may lead to reduced risk of delirium or chronic pain development. However, conclusive evidence on the effect of ketamine on pEEG indices is lacking and in particular, the effect of low dose ketamine on the NeuroSENSE monitor's WAVCNS index has not been investigated. This study will help to establish whether the WAVCNS index may be used as a reliable measure of clinical effect when one of two low doses of ketamine is used during general anesthesia. This is a significant step towards the development of a larger randomized controlled clinical trial in which the influence of ketamine on pEEG feedback-based anesthesia will be assessed.

Methods Study Design This randomized, open-label, feasibility study will be undertaken in a sample of healthy adult outpatient surgery patients under the direct and immediate supervision of an experienced anesthesiologist.

Intervention

Patients will undergo general anesthesia, consisting of continuous infusions of propofol (for anesthesia) and remifentanil (for analgesia). The study-specific intervention is the addition of EEG monitoring with the NeuroSENSE monitor in all three groups, and the addition of one of two possible ketamine doses (bolus and infusion) in two groups:

* Group 1: Ketamine 0.5 mg/kg loading dose followed by a 10 mcg/kg/min infusion
* Group 2: Ketamine 0.25 mg/kg loading dose followed by a 5 mcg/kg/min infusion
* Group 3: Control - No ketamine

Randomization Thirty study participants will be randomly allocated to one of three groups based on a randomization code assigned to them after they have provided their informed consent. Randomization will be performed in block sizes of six subjects to maintain relatively even group sizes throughout the study period.

Blinding The goal of this study is to integrate the protocol with an otherwise standard anesthetic. As a result, the anesthesiologist will be blinded to the NeuroSENSE monitor display, as the use of EEG monitoring is not currently part of standard practice. The anesthesiologist will instead rely on feedback from the other patient monitors in the OR, as they normally would. The NeuroSENSE monitor screen will be covered by an opaque card during the entire procedure, except for the displayed signal quality information. Blinding is required to avoid influencing the anesthesiologist's decisions based on EEG parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-54
* ASA I-II
* BMI 15-45
* Elective ACL repair surgery requiring general anesthesia, scheduled to take >60min
* Ability to read and understand the informed consent form

Exclusion Criteria

* Contraindications to ketamine use (e.g. severe cardiovascular disease, pacemaker, pheochromocytoma, malignant hypertension, intraocular pressure pathology, acute globe injury, hyperthyroidism)
* Contraindications to propofol (Anaphylactic reaction to eggs, egg products, soybeans or soy products)
* Contraindications to remifentanil (Hypersensitivity to fentanyl analogues)
* Known or suspected neurological disease (Tumor, stroke, neurodegenerative disease, major head injury; Abnormality in any previous EEG examination EEG (seizure disorder); Cognitive deficits (dementia, developmental delay))
* Acquired scalp or skull abnormalities
* Psychiatric illness (Severe depression, PTSD, psychosis; Any psychotropic medication taken in the past 7 days)
* History of drug misuse/abuse within past 30 days (Ketamine, cocaine, heroin, amphetamines, phencyclindine, lysergic acid (LSD), mescaline, psilocybin, Chronic alcoholism)
* Pre-operative sedative medication (e.g. midazolam) required
* Anticipated intra-operative or pre-operative use of nitrous oxide, catecholamines (dopamine, epinephrine, norepinephrine) or thyroid hormones
* Pregnant or nursing
* Currently enrolled in any other research study involving drugs or devices

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
WAVcns | Continually assessed throughout general anesthesia during thier surgery, approximately 1-2 hours.
  WAVcns is a measure of depth of hypnosis from the NeuroSENSE monitor.

SECONDARY OUTCOMES:
Total postoperative cumulative opioid requirements | During post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  All opioid medication will be recorded in the PACU. Will be calculated as morphine equivalent doses.
Occurrence and severity of pain | At least hourly during post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  Subjects report their pain intensity at rest and upon knee flexion, if possible, using a 0-10 numerical rating scale.
Post-operative nausea & vomiting (PONV) - Nausea | At least hourly during post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  Nausea is defined as the subjective report of upset stomach or urge to vomit, and will be measured using a self-reported numerical rating scale from 0 (no nausea) to 10 (the worst nausea imaginable) hourly or more frequently if needed. Standard nursing records will include any reports of post-operative nausea.
Post-operative nausea & vomiting (PONV) - Vomiting | At least hourly during post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  Vomiting is defined as the forcible ejection of stomach contents through the mouth. Standard nursing records will include any reports of post-operative vomiting.
Post-operative nausea & vomiting (PONV) - Retching | At least hourly during post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  Retching is defined as gastric and esophageal movements of vomiting without expulsion of vomitus. Standard nursing records will include any reports of post-operative retching.
Post-operative nausea & vomiting (PONV) - Anti-emetic medication | At least hourly during post-anesthesia care unit (PACU) stay, approximately 1-6 hours.
  Standard nursing records will include the dose and time of any anti-emetic medication given.
Postoperative shivering | Admission to post-anesthesia care unit (PACU), and 30 and 60 minutes thereafter during their PACU stay, approximately 1-6 hours.
  Shivering is based on a 4 point scale from 0 (no shivering) to 3 (Gross muscular activity involving the entire body)
Dreaming and awareness | Once subject is oriented to time, place, and person, in the post-anesthesia care unit (PACU). This questionnaire will take from 5-15 minutes to complete.
  A standard questionnaire will be administered.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Merchant, Principal Investigator — Fraser Health (Royal Columbian and Eagle Ridge Hospitals) and University of British Columbia
Locations (1):
- Fraser Health: Eagle Ridge Hospital, Port Moody, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Once data collection is complete, a de-identified version of the data may be made available to other researchers. This will be specifically stated in the consent form, and participants will be asked to provide their consent for releasing their anonymized data as well as for participating in the study. Participants may still participate in the study if they do not consent to make their data available.

REFERENCES:
- [Derived] van Heusden K, Cooke E, Brodie S, West N, Gorges M, Dumont GA, Ansermino JM, Merchant RN. Effect of ketamine on the NeuroSENSE WAVCNS during propofol anesthesia; a randomized feasibility trial. J Clin Monit Comput. 2021 May;35(3):557-567. doi: 10.1007/s10877-020-00511-0. Epub 2020 Apr 19. PMID 32307624